CLINICAL TRIAL: NCT06252324
Title: Sopravvivenza e Healing Rate di Due Tecniche di Otturazione Canalare: Studio Clinico Randomizzato
Brief Title: Success and Survival Rate of Tranmucosal Versus Bone Level Implants: Randomized Clinical Trial
Acronym: PERI-IMPLANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Fausto Zamparini, Fausto Zamparini, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 596-2022-SPER-AUSLBO
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- submerged implant placement with healing abtument (Experimental): the implant was placed flush to the bone crest after anaesthesia and with no flap elevation.
  A healing screw was positioned to have a transmucosal healing. the healing was removed after 3 months and cement restoration technique was performed in all cases.
  Interventions: Other: Prime taper implant + healing screw
- Tissue level implant placement cover screw (Other): the implant was placed above the bone crest after anaesthesia and with no flap elevation.
  A cover screw was positioned to have a tissue level healing. the screw was removed after 3 months and cement restoration technique was performed in all cases.
  Interventions: Other: Prime taper implant + cover screw

INTERVENTIONS:
Other: Prime taper implant + cover screw — tissue level implant placement with the addition of a cover screw
  Other Names: nonsubmerged healing
  Arms: Tissue level implant placement cover screw
Other: Prime taper implant + healing screw — bone level implant placement with the addition of a healing screw
  Other Names: submerged healing
  Arms: submerged implant placement with healing abtument

SUMMARY:
The purpose of this study is to assess changes in peri-implant tissues and the effectiveness of a tissue-level surgical technique. This technique will be compared with a bone-level surgical technique.

This is a post-marketing clinical investigation conducted in the Endodontics Department of the Dental Clinic at the University of Bologna. Patient recruitment and study conduction will follow the principles of the Declaration of Helsinki and adhere to major international guidelines (CONSORT).

Implants will be placed using either a bone-level or tissue-level surgical technique, corresponding to implants positioned at the level of the gingival mucosa or submerged implants, respectively. Randomization (1:1 ratio) will be conducted before surgery to create two treatment groups. The experimental group (Tissue Level) (n=40) consists of implants that will be placed with the exposed neck (Tissue-level surgical technique). The control group (n=40) comprises implants placed at the bone level (Bone-level surgical technique). The surgeon will be aware of patient assignment during the implant insertion procedures. The surgical procedure to uncover the implant neck (control group) will be performed 3 months after implant placement. The experimental group (Tissue Level technique) will not require a surgical intervention.

he following parameters will be assessed at 1, 6, 12, and 36 months after implant placement: Peri-implant parameters: Plaque score, Bleeding on Probing (BoP), and Papilla Index Radiographic parameters: Marginal Bone Level (MBL) Patient-Reported Outcome Measure (PROM): Post-operative pain (VAS) in the experimental group (non-submerged surgical technique) and the control group (submerged surgical technique).

DETAILED DESCRIPTION:
Objectives The purpose of this study is to assess changes in peri-implant tissues and the effectiveness of a tissue-level surgical technique. This technique will be compared with a bone-level surgical technique.

Materials and methods This is a post-marketing clinical investigation conducted in the Endodontics Department of the Dental Clinic at the University of Bologna. Patient recruitment and study conduction will follow the principles of the Declaration of Helsinki and adhere to major international guidelines (CONSORT).

The Endodontics Department has 10 dental units and typically sees 20-30 patients per day. Assuming an average of 1-2 patients per week meeting inclusion criteria, it is anticipated that at least 40 working weeks will be needed to achieve the minimum required sample. The recruitment period is estimated to be around 12-15 months to ensure the recruitment of the required number of patients. Participation in the study will be voluntary, contingent on obtaining written consent.

Implants will be placed using either a bone-level or tissue-level surgical technique, corresponding to implants positioned at the level of the gingival mucosa or submerged implants, respectively. Randomization (1:1 ratio) will be conducted before surgery to create two treatment groups. The experimental group (Tissue Level) (n=40) consists of implants that will be placed with the exposed neck (Tissue-level surgical technique). The control group (n=40) comprises implants placed at the bone level (Bone-level surgical technique). The surgeon will be aware of patient assignment during the implant insertion procedures. The surgical procedure to uncover the implant neck (control group) will be performed 3 months after implant placement. The experimental group (Tissue Level technique) will not require a surgical intervention.

Three months later, the impression will be taken using a digital scanner, and the custom titanium abutment will be secured within 15-21 days. A provisional single acrylic crown will be cemented with temporary cement as a temporary prosthetic rehabilitation. Thirty days later, a definitive prosthetic restoration will be applied using polycarboxylate cement.

All measurements and clinical/radiological evaluations will be performed by an operator who did not participate in the surgical and rehabilitative phases. The operator will be calibrated before conducting clinical evaluations. The following parameters will be assessed at 1, 6, 12, and 36 months after implant placement:

Peri-implant parameters: Plaque score, Bleeding on Probing (BoP), and Papilla Index Radiographic parameters: Marginal Bone Level (MBL) Patient-Reported Outcome Measure (PROM): Post-operative pain (VAS) in the experimental group (non-submerged surgical technique) and the control group (submerged surgical technique).

The plaque score will be evaluated at four sites (mesial, distal, buccal, and palatal) around the implant restorations and adjacent teeth. A dichotomous score will be assigned (0= no visible plaque at the soft margin; 1= visible plaque at the soft margin).

Bleeding on probing (BoP) will be measured at four sites (mesial, distal, buccal, and palatal) around the implant restorations and adjacent teeth. A dichotomous score will be assigned (0= no bleeding; 1= bleeding).

MBL will be evaluated on periapical radiographs of mesial and distal implant surfaces by measuring the distance between the implant platform reference point and the most coronal contact level between bone and implant using a scale divided into 0.1 mm steps. Evaluation endpoints are at 1, 3, 6, 12, and 36 months.

The Papilla Index will be measured in each rehabilitation: values 0 and 1 indicate absent or limited papilla growth, while values 2 and 3 indicate adequate papilla growth. Index 4 will indicate excessive papilla growth and hyperplasia. Evaluation endpoints are at 3, 6, and 36 months.

Post-operative pain will be assessed using the VAS scale, which includes 10 values representing the degree of pain (0= no pain, 10= maximum possible pain). The assessment will be conducted 3 months after implant placement, concurrently with the impression-taking procedures.

Sample Size The primary objective is the evaluation of peri-implant bone levels, which will be performed through the calculation of Marginal Bone Level (MBL). Sample size analysis was conducted using SigmaPlot software (version 13, Systat, Chicago, IL, USA). Assuming a confidence level of 90% and a margin of error of 15%, 25 patients per group (75 patients in total) will be required to detect a difference of approximately 20% between MBL values in the two groups. Considering a drop-out rate of about 10-15% during follow-up, 40 patients per group will be recruited (80 in total).

Data Management and Statistical Analysis

Data collected during the study will be recorded, processed, analyzed throughout the project, and stored in a pseudo-anonymous manner, along with the code identifying the Subject. Only authorized personnel will be able to link this code to the individual's identity. Data collected in Excel will be analyzed using SigmaPlot software. A Generalized Linear Model will be executed to assess any significant differences between the two groups at follow-ups (one month, three months, six months, twelve months, and thirty-six months) regarding different parameters (MBL, Plaque Score, BoP, and Papilla Index). Furthermore, a multiple linear regression with stepwise selection will be performed to analyze factors associated with MBL, Plaque Score, BoP, and Papilla Index.

Confidentiality of Collected Information

The data controller is the University of Bologna, and the responsible person is the Principal Investigator. Data resulting from the analyses will be processed with statistical methods to derive the information that constitutes the purpose of the research. The study manager and collaborators will have access to the data, bound by confidentiality and data processing obligations according to current regulations. Monitoring and verification personnel, the Ethics Committee, and Regulatory Authorities may directly access biological materials to verify study procedures and/or data to the extent allowed by current regulations. The study results will be the basis for a scientific publication, and even in this work, data will be reported anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years;
* Healthy or with mild functional limitations according to ASA classification 1-2 (16);
* Consumption of fewer than 10 cigarettes per day;
* Need for implant rehabilitation in a single-tooth edentulous area;
* Presence of adequate volumes of bone tissue (3.5mm thickness and 9mm height) to allow proper implant placement and optimal primary stability.

Exclusion Criteria:

* Age under 18 years;
* Medical and/or general contraindications to surgical procedures (ASA score ≥3) (16);
* Poor oral hygiene and lack of motivation and/or active clinical periodontal disease expressed by probing pocket depth >4 mm and bleeding on probing;
* Smoking more than 10 cigarettes per day;
* Systemic or local diseases that could compromise post-operative healing and osseointegration;
* Alcohol and/or drug abuse;
* Pregnancy or breastfeeding;
* Malocclusion and other occlusal disorders;
* Bisphosphonate therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Marginal bone level (MBL) around implants | immediately after implant insertion, 1 month, 3 months, 6 months, 12 months, 24 months and 36 months.
  analysis of bone level variations at different time frames
implant survival rate | 12 months, 24 months, 36 months from insertion
  number of implants still functional at the end of the follow-up

SECONDARY OUTCOMES:
post-operative pain | immediately after insertion, 3months after insertion (crown and abutment applications)
  analysis of post operative pain through Visual Analogical scale (VAS). The scale is constituted of 10 values. 0= no pain; 10=most intense pain

CONTACTS AND LOCATIONS:
Overall Officials: Maria Giovanna Gandolfi, Principal Investigator — Dibinem, University of Bologna
Locations (1):
- Endodontic clinical section, DIBINEM, UNiversity of Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided